CLINICAL TRIAL: NCT06069245
Title: The Acute Effects of Mitochondrial Antioxidant Supplementation on Metabolic Flexibility
Brief Title: MitoQ & Cardiopulmonary Responses During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ball State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1946841-3
Record Dates: First submitted 2023-09-25; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Healthy
MeSH Terms: interventions — mitoquinone

STUDY DESIGN:
Intervention Model Description: Double blind randomized placebo controlled crossover design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Gelatin capsules
  Interventions: Dietary Supplement: Placebo
- MitoQ (Experimental): Commercially available MitoQ (80mg)
  Interventions: Dietary Supplement: MitoQ

INTERVENTIONS:
Dietary Supplement: MitoQ — 80mg of MitoQ taken in one dose on one occasion.
  Arms: MitoQ
Dietary Supplement: Placebo — Gelatin capsules
  Arms: Placebo

SUMMARY:
Study Purpose: To examine the acute effects of antioxidant supplementation on energy use during a single bout of exercise in apparently healthy adult men and women.

Specifically this study examined the acute effect of MitoQ on:

1. cardiopulmonary responses to submax and maximal exercise
2. Energy expenditure and fat/carbohydrate oxidation during sub maximal exercise.

In a double-blind, randomized, placebo controlled, cross-over study design, participants performed 2 experimental trials which differed only in the supplement consumed (MitoQ or Placebo). Participants performed identical exercise protocols which consisted of a series of submaximal workloads followed by a ramp protocol to volitional exhaustion.

DETAILED DESCRIPTION:
Participants performed the following 3 study visits:

Visit 1 consisted of baseline resting measures including blood pressure and blood vessel health, blood biomarkers, and body composition assessments.

Visits 2 and 3 were the acute supplementation intervention(s) with either MitoQ or Placebo in a randomly designed order. These visits included an assessment of blood pressure and blood vessel health and an exercise test on a stationary cycle. There was a minimum of 48-72 hours between trials 2 and 3.

Visit 1

* Participants arrived at the laboratory fasted from all food and drink other than water for at least 12 hours. The following assessments were performed:
* Informed consent and health history questionnaire
* Resting heart rate, handgrip strength, and body composition
* Resting electrocardiogram (ECG)
* Blood biomarkers (Total cholesterol, HDL, LDL-C, and triglycerides as well as fasting blood glucose and HbA1c).
* Blood pressure

Visit 2 & 3 (performed in a randomized order differing only in the supplement consumed)

Acute supplementation intervention(s)

* The night before both the Placebo and MitoQ trials, participants were asked to eat the same meal at the same time of night and were provided with a standard Ensure shake to consume at 8:00pm the night before each trial.
* Upon arrival, they rested supine for ~10 minutes before consuming supplement (MitoQ or Placebo)
* Following consumption of the supplement or placebo, participants completed a graded aerobic exercise protocol. This test involved riding on a stationary cycle to exhaustion. The total test duration was ~30-45 minutes which included a break to rest between the submax and maximal portions. Heart function was monitored with an electrocardiogram (ECG). A gas analysis cart was used to determine the composition of the air breathed in and out during the test for the determination of substrate oxidation rates and VO2max. Heart rate was measured continuously throughout the exercise protocol from the ECG. Rate of perceived exertion (RPE) was measured every minute and blood pressure (BP) was performed every third minute of the exercise protocol. Additional measures of blood lactate via a finger stick were performed during the exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Be greater than or equal to 18 years of age
* Have a resting seated systolic blood pressure (SBP) of less than 160 mmHg and diastolic blood pressure (DBP) less than 100 mmHg
* Nonsmoker
* Body mass index (BMI) less than or equal to 35 kg/m2
* Considered physically inactive defined as participating in <150 min/week of moderate physical activity or <75 minutes/week of vigorous activity (ACSM).

Exclusion Criteria:

* participants that cannot complete the exercise protocol or have any signs/symptoms suggestive of cardiovascular or metabolic disease.
* Individuals that are currently on beta blockers
* diagnosed with type II diabetes will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | acutely (1 hr)
  VO2max

SECONDARY OUTCOMES:
Ventilation | acutely (1hr)
  L/min
Heart rate | acutely (1 hr)
  beats per minute
Blood pressure | acutely (1hr)
  mmHg
Maximal Fat Oxidation rate | acutely (1hr)
  g/min
Peak blood lactate | acutely (1hr)
  mmol

CONTACTS AND LOCATIONS:
Locations (1):
- Ball State University, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: No